CLINICAL TRIAL: NCT02224586
Title: Resting State Functional Magnetic Resonance Imaging Study of Jaundice Infants Before and After Light Treatment.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Ya-Fei Zhu, chief physician, Hangzhou Normal University
Other Study IDs: HNU_AH_jaundice fMRI
Record Dates: First submitted 2014-08-20; First posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Jaundice
MeSH Terms: conditions — Jaundice

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- light treatment: clinical routine treatment according to the doctor's advice
  Interventions: Device: light treatment

INTERVENTIONS:
Device: light treatment — clinical routine treatment according to the doctor's advice

SUMMARY:
It is just an observation study. The investigates want to explore the signal changes of resting state functional Magnetic resonance Imaging (fMRI) after light treatment in jaundice infants. Signal changes contain blood oxygenation level dependent (BOLD) and arterial spin labeling (ASL).Indicator of BOLD is amplitude of low-frequency fluctuation（ALFF).Indicator of ASL is cerebral blood flow (CBF).

The investigates assume that the children with jaundice after light therapy, ALFF and CBF will change. Focus on the globus pallidus and subthalamic nuclei. The two brain regions were proved to be abnormal in MRI T1, T2 structure signal in kernicterus.

Doctors observe the status of infants aside.Using monitoring probe can see clearly.

DETAILED DESCRIPTION:
resting state fMRI scan light therapy the second time resting state fMRI scan

ELIGIBILITY:
Inclusion Criteria:

* hyperbilirubinemia

Exclusion Criteria:

* asphyxia
* cerebral dysgenesis

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: municipal hospitals
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-03 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
amplitude of low-frequency fluctuation change before and after light treatment | before and after light treatment
  It is indicator of blood oxygenation level dependent.

SECONDARY OUTCOMES:
cerebral blood flow change before after light treatment | before and after light treatment
  It is indicator of arterial spin labeling.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Fei Zhu, Principal Investigator — Center for Cognition and Brain Disorders,Hangzhou Normal University
Locations (1):
- Center for Cognition and Brain Disorders, Hangzhou, Zhejiang, China